CLINICAL TRIAL: NCT06718413
Title: Quantifying and Treating Myofascial Dysfunction in Post Stroke Shoulder Pain
Brief Title: Myofascial Dysfunction in Post Stroke Shoulder Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00354872; 4R33AT012279-02 (NIH)
Record Dates: First submitted 2024-11-22; First posted 2024-12-05 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Hyaluronoglucosaminidase; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: study because each participant will receive both Human Recombinant Hyaluronidase and the placebo at some point during the study. For example, if the participant is assigned to receive the study drug for the first set of injections, the participant will receive placebo for the second set of injections.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Hyaluronidase plus saline (Treatment Arm) (Experimental): hyaluronidase plus saline injection
  Interventions: Drug: hyaluronidase plus saline
- Saline injection (Control Arm) (Experimental): normal saline injection
  Interventions: Drug: saline

INTERVENTIONS:
Drug: hyaluronidase plus saline — Injection of study drug with saline
  Other Names: Treatment Arm
  Arms: Hyaluronidase plus saline (Treatment Arm)
Drug: saline — injection of normal saline and no study drug
  Other Names: Control Arm
  Arms: Saline injection (Control Arm)

SUMMARY:
Shoulder pain is extremely common after stroke and occurs in 30-70% of patients. The pain may begin as early as one week after stroke, although peak onset and severity occurs around four months, and persists into the chronic stage. Chronic post stroke shoulder pain (PSSP) interferes with motor recovery, decreases quality of life, and contributes to depression. PSSP is thought to be caused mainly by damage to the myofascial tissues around the shoulder joint. Interestingly, an MRI study in patients with PSSP showed that the degree of structural damage to the muscles did not correlate with the degree of pain. Thus, the pathophysiology of myofascial dysfunction and pain in PSSP has not been elucidated leading to missed opportunities for early diagnosis and variable success with pain management.

The accumulation of hyaluronic acid (HA) in muscle and its fascia can cause myofascial dysfunction. HA is a glycosaminoglycan (GAG) consisting of long-chain polymers of disaccharide units of glucuronic acid and N-acetylglucosamine and is a chief constituent of the extracellular matrix of muscle. In physiologic quantities, HA functions as a lubricant and a viscoelastic shock absorber, enabling force transmission during contraction and stretch. Reduced joint mobility and spasticity result in focal accumulation and alteration of HA in muscle. This can lead to the development of stiff areas and taut bands, dysfunctional gliding of deep fascia and muscle layers, reduced range of motion (ROM), and pain. However, the association of muscle HA accumulation with PSSP has not been established.

The investigators have quantified the concentration of HA in muscle using T1rho (T1ρ) MRI and found that T1ρ relaxation time is increased in post stroke shoulder pain and stiffness. Furthermore, dynamic US imaging using shear strain mapping can quantify dysfunctional gliding of muscle that may generate pain during ROM. Myofascial dysfunction can result in non-painful reduction in ROM (latent PSSP), which may become painful due to episodic overuse injury producing greater shear dysfunction (active PSSP). Hence, shear strain mapping may differentiate between latent versus active PSSP. Thus, quantitative Motor Recovery (MR) and US imaging may serve as useful biomarkers to elucidate the pathophysiology of myofascial dysfunction.

DETAILED DESCRIPTION:
Aim 1: Quantify the extent of HA accumulation in shoulder muscles using T1rho MRI before and after treatment with hyaluronidase injections versus placebo in patients with PSSP. Hypothesis: The primary objective will be to demonstrate that dysfunctional shoulder girdle muscles on the paretic side in patients with PSSP will show decreased T1ρ relaxation times in the infraspinatus muscle after treatment with hyaluronidase injections compared with placebo 5-7 weeks post-injection.

Aim 2. Determine maximum sheer strain in shoulder muscles using US shear strain mapping before and after treatment with hyaluronidase injections versus placebo in patients with PSSP. Research Hypothesis: Shear strain on the paretic side in patients with PSSP measured using ultrasound shear mobility between the pectoralis major and minor muscles will decrease after treatment with hyaluronidase injections compared with placebo 5-7 weeks post-injection.

Aim 3. Assess the impact of hyaluronidase injections compared with placebo on shoulder pain, pain free range of motion, upper limb motor impairment, function and quality of life in patients with PSSP. Hypothesis: Hyaluronidase injections compared with placebo in patients with PSSP will lead to (1) reduced pain as assessed using the pain questionnaires and lower pain-pressure thresholds with quantitative sensory testing using an algometer; (2) increased pain free range of motion in most affected shoulder joints; (3) reduced upper limb motor impairment measured using the Fugl-Meyer Scale; (4) increased function measured using the Wolf Motor Function Test; and (5) improved quality of life measured using the Stroke Specific Quality of Life scale.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years;
* hemiparesis from an ischemic or hemorrhagic stroke;
* time since cerebral injury 3-180 months prior;
* show a difference of more than 10 degrees of passive ER-ROM between non-paretic and paretic shoulders with or without pain
* ability to give informed consent and HIPAA authorization, and comply with study protocols;

Exclusion Criteria:

* treatment of spasticity with Botulinum toxin or intrathecal baclofen within the past three months, phenol injections within the past 12 months, or ongoing adjustment of anti-spastic medications;
* other neurologic condition that may affect motor response (e.g., Parkinson's disease, Amyotrophic Lateral Sclerosis (ALS), MS);
* clinically significant cognitive dysfunction with score <19 on Folstein's Mini Mental Status Examination or positive depression screening on the Patient Health Questionnaire (PHQ)-9;
* pregnancy;
* known hypersensitivity to hyaluronidase;
* standard contraindications for MRI;
* have non-musculoskeletal PSSP such as only central pain or chronic regional pain syndrome (CRPS)
* any condition that will preclude the patient from completing the protocol as determined by the PI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
T1ρ relaxation times (ms) in the treatment group | Baseline, up to 7 weeks post first injection
  Aim 1: T1ρ relaxation times in the treatment group. The primary endpoint will be change in T1ρ relaxation times on MRI in the shoulder girdle muscles of the paretic side between the baseline visit and 5-7 weeks post-first injection (i.e., post injection follow up at Visit 5/ end of Phase 1).

SECONDARY OUTCOMES:
Ultrasound shear strain | 7 weeks
  Percent shear strain obtained via ultrasound in the two groups. Higher shear strain is better.
Pain rating as assessed by algometer | 7 weeks
  Pain rating on quantitative sensory testing of shoulder muscles. Lower pain rating is better.
Pain free range of motion | 7 weeks
  Range of motion for the most affected shoulder movement. Higher range of motion is better.
Upper limb motion impairment as assessed by the Fugl-Meyer Scale | 7 weeks
  Upper limb Fugl-Meyer scale; score range 0-66 with higher numbers reflecting less arm impairment
Upper limb function as assessed by Wolf Motor Function Test (time) | 7 weeks
  Participants are given a battery of functional tasks that are timed and scored on movement quality. Score range is 0-120, lower scores being better.
Quality of life as assessed by the Stroke Impact Scale | 7 weeks
  Scores range from 0-100, with higher score showing better quality of life and lower stroke impact.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Cao, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No